CLINICAL TRIAL: NCT07251101
Title: A Randomized, Parallel, Open-label With Blinded Assessment Study Comparing Hemodynamic Profiles Between Remimazolam- and Propofol-based Total Intravenous Anesthesia in Patients Undergoing Robot-assisted Gynecologic Surgery
Brief Title: Hemodynamic Effects of Remimazolam vs Propofol During Robot-assisted Gynecologic Surgery
Acronym: By_HD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ilsan Cha hospital (Other)
Responsible Party: Principal Investigator, Joohyun Lee, Assistant Professor, Department of Anesthesiology and Pain Medicine, CHA University, Ilsan Cha hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ICHA 2025-07-005
Record Dates: First submitted 2025-09-25; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia, Intravenous; Hemodynamic Stability; Gynecologic Surgery
Keywords: remimazolam; propofol; hemodynamics; laparoscopic surgery; general anesthesia; Trendelenburg position; pneumoperitoneum; gynecologic surgery; total intravenous anesthesia (TIVA)
MeSH Terms: conditions — Pneumoperitoneum | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group_R (Experimental): TIVA with remimazolam plus remifentanil
  Interventions: Drug: Remimazolam
- Group_P (Active Comparator): TIVA with propofol plus remifentanil
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Induction with remimazolam 6 mg·kg-¹·h-¹ with remifentanil Ce 4 ng·mL-¹ (Minto model); maintenance remimazolam 1-2 mg·kg-¹·h-¹, titrated (±0.2) to maintain PSI 25-50 and hemodynamic targets. Standard care otherwise per protocol.
  Other Names: Byfavo
  Arms: Group_R
Drug: Propofol — Induction with propofol Ce 4 ng·mL-¹ with remifentanil Ce 4 ng·mL-¹; maintenance propofol Ce 2.5-3.5 ng·mL-¹, titrated (±0.2) to maintain PSI 25-50 and hemodynamic targets. Standard care otherwise per protocol.
  Other Names: Fresofol MCT 2%
  Arms: Group_P

SUMMARY:
This single-center study at CHA Ilsan Medical Center compares intraoperative hemodynamics between remimazolam- and propofol-based total intravenous anesthesia (TIVA) in patients undergoing robot-assisted gynecologic surgery requiring pneumoperitoneum and steep Trendelenburg positioning.

DETAILED DESCRIPTION:
This study aims to compare intraoperative hemodynamic characteristics between remimazolam- and propofol-based total intravenous anesthesia (TIVA) in patients undergoing robot-assisted gynecologic surgery. Continuous invasive blood pressurewill be analyzed to evaluate time-weighted average (TWA) and area-under-the-curve (AUC) differences between groups. The study is designed as a randomized, parallel, open-label with blinded assessment trial.

ELIGIBILITY:
Inclusion Criteria:

* Female patients <65 years of age
* American Society of Anesthesiologists (ASA) physical status I-II
* Scheduled to undergo robotic hysterectomy under general anesthesia

Exclusion Criteria:

* Body mass index (BMI) > 35 kg/m²
* Baseline hypotension (systolic blood pressure <100 mmHg) or bradycardia (heart rate <60 bpm)
* History of ischemic heart disease or cardiac conduction block
* Significant cardiopulmonary disease, including hypoxemia (SpO₂ <90%), uncontrolled asthma, or chronic obstructive pulmonary disease (COPD)
* Use of inhalational anesthetics during anesthesia
* Conversion from robotic/laparoscopic surgery to open laparotomy

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
MAP (Time-Weighted Average) | From induction start (first anesthetic administration) to operating room exit (transfer from OR), approximately up to 5 hours per participant.
  Continuous invasive arterial pressure is recorded throughout anesthesia. For each participant, TWA-MAP is computed as the integral of MAP over elapsed time divided by total observation time (trapezoidal rule). Data are aggregated at ~1-min resolution when possible. Implausible artifacts (e.g., MAP <30 or >180 mmHg) are excluded. The primary comparison is the between-group difference in TWA-MAP (Remimazolam vs Propofol) for validating hypothesis(remimazolam-based TIVA maintains ≥20% higher intraoperative MAP than Propofol-based TIVA). Primary analysis will use ANCOVA adjusting for baseline MAP and prespecified covariates, with a one-sided significance level of 0.05.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) for Hypertensive Burden | From anesthesia induction to operating room exit, assessed continuously during surgery (approximately 2 to 5 hours per participant).
  Continuous invasive arterial pressure is recorded throughout anesthesia. For each participant, the AUC above the hypertensive threshold (SBP ≥140 mmHg or MAP ≥100 mmHg) is calculated as mmHg·minutes using the trapezoidal rule. This measure represents the cumulative burden of intraoperative hypertension. Group comparisons will assess whether remimazolam-based TIVA differs from propofol-based TIVA in hypertensive burden.
Area Under the Curve (AUC) for Hypotensive Burden | From anesthesia induction to operating room exit, assessed continuously during surgery (approximately 2 to 5 hours per participant).
  Continuous invasive arterial pressure is recorded throughout anesthesia. For each participant, the AUC below the hypotensive threshold (SBP <90 mmHg or MAP <65 mmHg) is calculated as mmHg·minutes using the trapezoidal rule. This measure represents the cumulative burden of intraoperative hypotension. Group comparisons will assess whether remimazolam-based TIVA differs from propofol-based TIVA in hypotensive burden.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - CHA Ilsan Medical Center, Goyang-si, Gyeonggi-do
  - CHA Ilsan Medical Center, Goyang-si

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Summary results will be published in peer-reviewed journals and presented at scientific meetings.